CLINICAL TRIAL: NCT07341607
Title: Effect of Structured Patient Education on Anxiety Levels and Quality of Life in Patients Undergoing Extracorporeal Shock Wave Lithotripsy: A Randomized Controlled Trial
Brief Title: STRUCTURED PATIENT EDUCATION IN ESWL PATIENTS
Acronym: ESWL-EDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Cemile Nida Kayış, Lecturer, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ESWL-EDU-RCT-2025
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Urolithiasis; ESWL
Keywords: Urolithiasis; Patient Education; Quality of Life; Anxiety; Nurse's Role; Nursing Care
MeSH Terms: conditions — Urolithiasis; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A total of 188 eligible patients will be enrolled in the study. Participants will be randomly assigned to the intervention or control group using permuted block randomization with a block size of four, resulting in two groups of 94 patients each. Randomization will be conducted by an independent researcher not involved in other study procedures.
  The researcher delivering the intervention will not be blinded, whereas outcome assessors will be blinded to group allocation. Accordingly, the study is designed as a single-blind randomized controlled trial.
  Control Group Standard patient information Intervention Group Participants in the intervention group will receive a nurse-led structured patient education program covering the pre- and post-ESWL periods. The program is based on current European Association of Urology and American Urological Association guidelines and relevant scientific literature.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Standard Patient Information (No Intervention)
- Intervention Group - Nurse-Led Structured Patient Education (Experimental): Intervention Group - Nurse-Led Structured Patient Education
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — Intervention Group Patients in the intervention group will receive a nurse-led structured patient education program covering both the pre- and post-extracorporeal shock wave lithotripsy (ESWL) periods. The education program has been developed in accordance with the current urolithiasis guidelines published by the European Association of Urology (Skolarikos et al., 2025) and the American Urological Association (Akram et al., 2024), as well as relevant up-to-date scientific literature (Geraghty et al., 2023; Jiang et al., 2021; Kasab et al., 2023; Koudonas et al., 2025; Tzelves et al., 2021).
  Arms: Intervention Group - Nurse-Led Structured Patient Education

SUMMARY:
Urolithiasis is a common urological disease with an increasing prevalence and high recurrence rates, negatively affecting patients' quality of life. Extracorporeal shock wave lithotripsy is a frequently preferred non-invasive treatment option in appropriate cases; however, uncertainties related to the procedural process and inadequate patient information may lead to increased anxiety and a decline in quality of life. Structured patient education delivered under nurse leadership has emerged as a potential approach to mitigate these adverse effects. Nevertheless, studies evaluating the impact of structured patient education on anxiety levels and quality of life in patients undergoing extracorporeal shock wave lithotripsy remain limited.

ELIGIBILITY:
Inclusion Criteria:

Aged between 18 and 65 years, Diagnosed with urolithiasis, Scheduled for elective extracorporeal shock wave lithotripsy (ESWL), Undergoing ESWL for the first time.

Exclusion Criteria:

Previous history of ESWL treatment, Urolithiasis cases requiring urgent intervention, Presence of renal insufficiency, active urinary tract infection, coagulopathy, or severe cardiopulmonary comorbidities, Inability to discontinue anticoagulant or antiplatelet therapy, Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: | Baseline (pre-procedure) and 4 weeks after discharge
  Change in quality of life assessed by the SF-12 Physical and Mental Component Summary scores from baseline (pre-procedure) to 4 weeks after discharge.

SECONDARY OUTCOMES:
Secondary Outcome: | Baseline (pre-procedure) and 4 weeks after discharge
  Change in anxiety levels assessed by the State-Trait Anxiety Inventory (STAI-I and STAI-II) from baseline to 4 weeks after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Cemile Nida Kayış, Principal Investigator — KTO Karatay University
Locations (1):
- Konya City Hospital, Department of Urology, Konya, Lecturer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data collected in this study will not be shared with other researchers in order to protect participant confidentiality and comply with data protection regulations. The data will be accessed only by the research team and will be analyzed in an anonymized manner. Study findings will be reported at an aggregate level, and no individual-level data will be made publicly available.

REFERENCES:
- [Result] Skolarikos A, Geraghty R, Somani B, Tailly T, Jung H, Neisius A, Petrik A, Kamphuis GM, Davis N, Bezuidenhout C, Lardas M, Gambaro G, Sayer JA, Lombardo R, Tzelves L. European Association of Urology Guidelines on the Diagnosis and Treatment of Urolithiasis. Eur Urol. 2025 Jul;88(1):64-75. doi: 10.1016/j.eururo.2025.03.011. Epub 2025 Apr 22. PMID 40268592
- See also: Related Info — https://journals.lww.com/jehp/fulltext/2024/11290/the_effect_of_education_on_pre_operative_anxiety.445.aspx